CLINICAL TRIAL: NCT02677077
Title: MRI and Clinical Disease Activity in Patients Treated Long Term With Natalizumab
Brief Title: Clinical Disease Activity With Long Term Natalizumab Treatment
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: BEL-TYS-14-10727
Record Dates: First submitted 2015-12-03; First posted 2016-02-09 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: RRMS; MRI
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Czech Republic: Approximately 230 participants with RRMS receiving commercial natalizumab in Czech Republic
  Interventions: Drug: natalizumab
- Belgium: Approximately 70 participants with RRMS receiving commercial natalizumab in Belgium
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — Participants with RRMS receiving commercial natalizumab in Belgium and Czech Republic
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of the study is to retrospectively investigate the proportion of participants free of new or enlarging fluid-attenuated inversion recovery (FLAIR) lesions over time in approximately 300 Relapsing-Remitting Multiple Sclerosis (RRMS) participants with regular MRI follow-up, who have received natalizumab ≥24 month from two different observational cohorts: 1) approximately 230 participants from the Czech Republic; and 2) approximately 70 participants from Belgium. The secondary objectives of this study are as follows: Brain volume change by various measures; Changes in the number and volume of magnetic resonance imaging (MRI) lesions; No evidence of disease activity (NEDA) with and without brain volume change.

DETAILED DESCRIPTION:
Natalizumab will not be provided to participants by Biogen as a part of this study. Participants will remain on natalizumab therapy as prescribed by their physician.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RRMS.
* Continuous treatment with natalizumab of ≥24 months. In case of a treatment interruption from natalizumab ≥60 days after a total treatment period of ≥24 months, only the treatment prior to the interruption will be analyzed. Any data after this treatment interruption (even if the patient restarts natalizumab) will not be analyzed/collected.
* ≥1 MRI scan of sufficient quality for reliable measurement.
* Baseline MRI scan ≤6 month prior to natalizumab treatment acquired.
* ≥1 MRI scan of sufficient quality for reliable measurement taken while on natalizumab treatment for ≥6 months.
* EDSS ≤ 6.5.

Key Exclusion Criteria:

* Anti-natalizumab antibody detection.
* Prior treatment with alemtuzumab.
* Prior treatment with mitoxantrone within 12 months of the first infusion of natalizumab.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been receiving treatment with natalizumab for ≥24 months.
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
Change over time in the number of participants free of new or enlarging FLAIR lesions | Treatment years 3 and 4
  Lesions that are ≥5 mm per scan (slice thickness 3 mm) as assessed by semiautomatic lesion count (by the Icometrix algorithm).

SECONDARY OUTCOMES:
Annualized brain volume change rate as assessed by % change in brain parenchymal fraction [BPF] | Post long term treatment with natalizumab (>2 years) through Year 4
Annualized brain volume change rate as assessed by percent brain volume change [PBVC] | Post long term treatment with natalizumab (>2 years) through Year 4
Annualized brain volume change rate as assessed by white matter [WM] and gray matter [GM] atrophy) | Post long term treatment with natalizumab (>2 years) through Year 4
Cumulative number of new ≥6-month confirmed T1-hypointense lesions | Post long term treatment with natalizumab (>2 years) through Year 4
Annualized T1-hypointense and FLAIR lesion volume change | Post long term treatment with natalizumab (>2 years) through Year 4
Cumulative percent change in T1-hypointense and FLAIR lesion volume | Post long term treatment with natalizumab (>2 years) through Year 4
Cumulative number of ≥6-month-confirmed T1-hypointense lesions arising from new on- treatment Gadolinium (Gd+)-enhancing lesions | Post long term treatment with natalizumab (>2 years) through Year 4
  No relapse and no ≥6-month confirmed Expanded Disability Status Scale (EDSS) progression and no new or enlarging FLAIR lesions and no new Gd+-enhancing lesions
Number of total participants and 4-year completers with NEDA as measured by clinical measures | Post long term treatment with natalizumab (>2 years) through Year 4
  No relapse and no ≥6-month confirmed EDSS progression and no new or enlarging FLAIR lesions and no new Gd+-enhancing lesions, brain volume change rate as assessed by PBVC
Number of total participants and 4-year completers with NEDA as measured by radiological measures | Post long term treatment with natalizumab (>2 years) through Year 4
  No new or enlarging FLAIR lesions and no new Gd+-enhancing lesions
Number of participants with brain volume loss ≤0.2% and ≤0.4% | Post long term treatment with natalizumab (>2 years) through Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- Belgium (3):
  - Research Site 1, Brussels
  - Research Site 2, Brussels
  - Research Site, Overpelt
- Research Site, Prague, Czechia